CLINICAL TRIAL: NCT04613557
Title: Open-label Phase I, Multi-center Study to Determine the Recommended Dose of CYAD-211 After a Non-myeloablative Preconditioning Chemotherapy in Multiple Myeloma Patients With Relapsed or Refractory Disease
Brief Title: Safety, Activity and Cell Kinetics of CYAD-211 in Patients With Relapsed or Refractory Multiple Myeloma
Acronym: IMMUNICY-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-211-001
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-06

CONDITIONS: Relapse/Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Cyclophosphamide; fludarabine phosphate; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CYAD-211 (Experimental): Infusion post preconditioning non-myeloablative chemotherapy
  Interventions: Biological: CYAD-211; Drug: Endoxan; Drug: Fludara

INTERVENTIONS:
Biological: CYAD-211 — Allogeneic anti-BCMA chimeric antigen receptor (CAR) T-cell
Drug: Endoxan — Preconditioning chemotherapy
  Other Names: cyclophosphamide
Drug: Fludara — Preconditioning chemotherapy
  Other Names: Fludarabine

SUMMARY:
The purpose of the IMMUNICY-1 study is to assess the safety, activity and cell kinetics of CYAD-211 in adults with relapsed or refractory multiple myeloma after a lymphodepletion regimen with fludarabine and/or cyclophosphamide

DETAILED DESCRIPTION:
This study aims to determine the recommended dose of the allogeneic CYAD-211 (anti-BCMA CAR-T) cells after a non-myeloablative preconditioning chemotherapy in multiple myeloma (MM) patients with relapsed or refractory disease.

ELIGIBILITY:
1. Documented diagnosis of MM with relapsed or refractory disease to at least two prior MM treatment regimens which should include exposure to IMiD and PIs either alone or in combination.
2. Presence of measurable disease as per International Myeloma Working Group (IMWG) Response Criteria
3. Eastern Cooperative Oncology Group (ECOG) below or equal 2
4. Adequate hematologic, renal, hepatic, pulmonary, and cardiac function

Exclusion Criteria:

1. History or presence of clinically relevant central nervous system (CNS) tumor involvement.
2. Autologous stem cell transplant within 12 weeks of registration or an allogeneic stem cell transplant within 6 months of starting study treatment.
3. Any investigational agent within 3 weeks prior to the initiation of the non-myeloablative preconditioning chemotherapy).
4. Prior systemic therapy for MM within 14 days prior to the initiation of the non-myeloablative preconditioning chemotherapy.
5. Prior treatment with any BCMA-targeted therapy and which has not achieved at least a partial response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2037-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities | Up to 36 days post-infusion.
  Occurrence of Dose Limiting Toxicities

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Nyu Langone Hospitals, New York, New York
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Institut Jules Bordet, Brussels
  - AZ DELTA, Roeselare